CLINICAL TRIAL: NCT01420952
Title: PET Imaging of Brain mGlu1 Receptors Using [11]LY2428703
Brief Title: Imaging of Brain Receptors Using (11C)mGlu1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 110229; 11-M-0229
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2012-11-27

CONDITIONS: Dosimetry; Pharmacokinetics
Keywords: Positron Emission Tomograhy (PET); Metabolic Glutamate Receptors; Brain

INTERVENTIONS:
Drug: [11C]LY2428703

SUMMARY:
Background:

- (11C)mGlu1 is a new drug that helps to show where a protein, mGluR1, is found in the brain. The drug contains a small amount of radioactivity that can be detected by imaging studies like positron emission tomography (PET) scans. By looking at the mGluR1 receptors, researchers hope to better understand how they are involved in general health, brain disorders, and addiction.

Objectives:

* To test how (11C)mGlu1 is distributed in the brain and body.
* To measure how mGluR1 receptors display (11C)mGlu1 during imaging studies.

Eligibility:

- Healthy volunteers between 18 and 50 years of age.

Design:

* Participants will be screened with a medical history, physical exam, and blood and urine tests. This study requires four visits to the NIH Clinical Center.
* Participants will have an initial evaluation, a magnetic resonance imaging (MRI) scan, a PET scan, and a final blood sample after the PET scan, all at different visits.
* The MRI and PET scans will focus on the brain. Participants will receive (11C)mGlu1, and have scans to see how it shows up in the brain.
* Some participants will have whole body imaging studies to see how (11C)mGlu1 shows up in the body.

DETAILED DESCRIPTION:
Metabotropic glutamate receptors (mGluRs) are G-protein coupled receptors that respond to glutamate by activating proteins inside nerve cells that affect cell metabolism, thereby fine-tuning the signals sent between cells to maintain balance in neuronal activity. mGluR receptor subtype 1 (mGluR1s) are located in several brain regions, including the cerebellum, hippocampus, olfactory bulb, and basal ganglia. mGluR1 activation stimulates phospholipase C, resulting in phosphoinositide hydrolysis and increased intracellular Ca(2+) levels. Detailed study of mGluR1s has heretofore been hindered by the lack of high affinity and of selective ligands for this receptor subtype.

The present protocol will use a new PET ligand [C(11)]mGlu1 to 1) perform kinetic brain imaging to quantify mGluR1 binding parameters in brain and determine the reliability and reproducibility of these measures in 15 healthy volunteers (Phase 1); and 2) if the tracer proves successful in Phase 1, we will estimate radiation-absorbed doses of [C(11)]mGlu1 in healthy human subjects by performing whole body imaging (Phase 2).

Successful development of a PET ligand to image mGlurR1 would have a strong impact on clinical management of brain disorders characterized by disruptions in glutamatergic transmission, including anxiety and stress disorders, drug addiction, epilepsy, Huntington s disease, and Parkinson s disease.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy volunteers subjects aged 18 50 with medical history/physical exam, electrocardiogram (ECG), and laboratory tests within normal limits within 60 days of the PET scan.

EXCLUSION CRITERIA:<TAB>

* <TAB>Lifetime psychiatric illness or severe systemic disease based on history and physical exam.
* <TAB>Serious medical illness likely to modify brain anatomy and/or physiology (seizure disorders, past brain surgery, etc.)
* <TAB>High blood pressure, as demonstrated by at least two resting measurements above 140/100, separated by at least 30 min.
* <TAB>Any current substance or alcohol abuse, with the exception of nicotine.
* <TAB>Positive urine toxicology screen
* <TAB>Radiation exposure from participation in other research protocols or clinical care in the last year such that the additional radiation exposure from this protocol would exceed annual limits.
* <TAB>Pregnancy or breastfeeding.
* <TAB>Claustrophobia (Part 1 only).
* <TAB>metallic (ferromagnetic) implants, including pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, shrapnel fragments, and possible small metal fragments in the eye (Part 1 only).
* <TAB>Unable to lie flat on back for up to 2.5 hours.
* <TAB>Positive HIV test.
* <TAB>Inability to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-07-29; Primary Completion 2012-11-27 (Actual); Study Completion 2012-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kunishima N, Shimada Y, Tsuji Y, Sato T, Yamamoto M, Kumasaka T, Nakanishi S, Jingami H, Morikawa K. Structural basis of glutamate recognition by a dimeric metabotropic glutamate receptor. Nature. 2000 Oct 26;407(6807):971-7. doi: 10.1038/35039564. PMID 11069170
- [Background] Conn PJ, Pin JP. Pharmacology and functions of metabotropic glutamate receptors. Annu Rev Pharmacol Toxicol. 1997;37:205-37. doi: 10.1146/annurev.pharmtox.37.1.205. PMID 9131252
- [Background] Spooren W, Ballard T, Gasparini F, Amalric M, Mutel V, Schreiber R. Insight into the function of Group I and Group II metabotropic glutamate (mGlu) receptors: behavioural characterization and implications for the treatment of CNS disorders. Behav Pharmacol. 2003 Jul;14(4):257-77. doi: 10.1097/01.fbp.0000081783.35927.8f. PMID 12838033